CLINICAL TRIAL: NCT02149394
Title: Efficacy of Ice Popsicle in the Management of Thirst in the Immediate Postoperative Period: Randomized Clinical Trial
Brief Title: Ice Popsicle for Thirst Relief of the Surgical Patient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Estadual de Londrina (Other)
Responsible Party: Principal Investigator, Marilia Ferrari Conchon, Master of science degree in nursing, Universidade Estadual de Londrina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16707313.5.0000.5231
Record Dates: First submitted 2014-05-17; First posted 2014-05-29 (Estimated); Last update posted 2014-05-29 (Estimated); Status verified 2014-05

CONDITIONS: Thirst
Keywords: Thirst; Ice; Water; Perioperative Nursing; Recovery Room

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ice (Experimental): The concealment of allocation was performed through the use of individual opaque envelopes numbered externally in sequence, containing information of the group randomly defined. This step was carried out by a researcher who did not take part in data collection.Thirst intensity was measured within the range from 1 to 10 according to the numeric visual analogue scale.The experimental group received an ice popsicle made of 10 mL mineral water.The ice popsicles were made according to the predetermined volumes and packed in the freezer of the anesthetic recovery room at the institution researched. The block of ice was supported by a stick, allowing the patients to control the intensity of cold conferred by the ice for their comfort.
  Interventions: Other: Ice popsicle
- Water (Active Comparator): The concealment of allocation was performed through the use of individual opaque envelopes numbered externally in sequence, containing information of the group randomly defined. This step was carried out by a researcher who did not take part in data collection.Thirst intensity was measured within the range from 1 to 10 according to the numeric visual analogue scale. The usual activities adopted by the nursing staff of the anesthetic recovery room were maintained for the control group that received 10 mL mineral water at room temperature in a syringe.
  Interventions: Other: Water at room temperature

INTERVENTIONS:
Other: Ice popsicle — Patients were assessed according to the following criteria before each intervention: level of awareness; airway protection capacity; and absence of nausea and vomiting, according to the Safety Protocol for Thirst Management. The experimental group received an ice popsicle made of 10 mL mineral water.
  The ice popsicles were made according to the predetermined volumes and packed in the freezer of the anesthetic recovery room at the institution researched. The block of ice were supported by a stick, allowing the patients to control the intensity of cold conferred by the ice for their comfort.
  Arms: Ice
Other: Water at room temperature — Patients were assessed according to the following criteria before each intervention: level of awareness; airway protection capacity; and absence of nausea and vomiting, according to the Safety Protocol for Thirst Management. The usual activities adopted by the nursing staff of the anesthetic recovery room were maintained for the control group that received 10 mL mineral water at room temperature in a syringe.
  Arms: Water

SUMMARY:
The purpose of this study is to assess the efficacy of ice popsicle compared with water at room temperature in relieving thirst in the immediate postoperative period . The hypothesis of the study is that ice has 20% greater efficacy than water to relieve thirst in the immediate postoperative period.

DETAILED DESCRIPTION:
There is evidence that ice is effective in relieving thirst in surgical patients, because, by stimulating the oral receptors sensitive to cold, ice decreases the need to ingest large volumes of liquids to satisfy thirst. This way, the risk of bronchoaspiration due to gastric fullness is avoided and discomfort with dry mouth is reduced. Preliminary evidence, therefore, indicates that the use of ice chips have greater efficacy than water at room temperature in relieving thirst. However, there is no scientific evidence from controlled studies with results that can be generalized with respect to a safe volume and adequate frequency of ice administered to reduce thirst in the immediate postoperative period.Considering that the gold standard for the study of a symptom is based on individuals' perceptions and their reports, this study is justified in order to assess the effectiveness of ice compared with water at room temperature in relieving thirst in the immediate postoperative period.

ELIGIBILITY:
Inclusion Criteria:

* aged between 18 and 65 years;
* undergoing more than eight-hour preoperative fasting;
* expressing thirst spontaneously or stimulated with intensity greater than or equal to three according to the numeric visual analogue scale;
* receiving opioids or anticholinergics during surgery;
* duration of anesthesia exceeding one hour;
* having been approved in the assessment by the Safety Protocol of Thirst Management;
* signing the informed consent during the preoperative period.

Exclusion Criteria:

* patients who had intake or swallowing restrictions.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2013-08; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Change in the intensity of the final thirst assessment with respect to the initial thirst assessment. | 1 hour
  5 evaluations of thirst intensity every 15 minutes during the first hour postoperatively.
  Thirst intensity was measured within the range from 1 to 10 in 1.0 intervals as reported by patients when orally required "how thirsty are you now?"according to the visual analogue scale. Zero means not thirsty at all and ten the worst thirst sensation that the patient have ever had.

SECONDARY OUTCOMES:
Reaching the point of satiety over one-hour assessment presented by the experimental and control groups. | 1 hour
  5 evaluations of thirst intensity and satiety every 15 minutes during the first hour postoperatively. Thirst intensity was measured within the range from 1 to 10 in 1.0 intervals as reported by patients when orally required "how thirsty are you now?"according to the visual analogue scale. Zero means not thirsty at all and ten the worst thirst sensation that the patient have ever had.according to the visual analogue scale. Satiety was characterized as intensity of thirst = zero (0).

CONTACTS AND LOCATIONS:
Overall Officials: Marilia F Conchon, Principal Investigator — Universidade Estadual de Londrina; Ligia F Fonseca, PhD, Study Director — Universidade Estadual de Londrina
Locations (1):
- University hospital - State University of Londrina, Londrina, Paraná, Brazil